CLINICAL TRIAL: NCT01970007
Title: Evaluation of the Zilver® Vena™ Venous Stent in the Treatment of Symptomatic Iliofemoral Venous Outflow Obstruction
Brief Title: VIVO Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-010
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Symptomatic Venous Outflow Obstruction in the Iliofemoral Vein
Keywords: venous; outflow obstruction; iliofemoral vein

ARMS (1):
- Zilver Vena Venous Self-Expanding Stent (Experimental)
  Interventions: Device: Zilver Vena Venous Self-Expanding Stent

INTERVENTIONS:
Device: Zilver Vena Venous Self-Expanding Stent — stenting
  Other Names: venous stent

SUMMARY:
The purpose of the VIVO Clinical Study is to evaluate the safety and effectiveness of the Zilver® Vena™ Venous Stent in the treatment of symptomatic iliofemoral venous outflow obstruction.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic venous outflow obstruction in one iliofemoral venous segment (i.e., one limb) per patient, demonstrated by:

  * CEAP "C" ≥ 3, or
  * VCSS pain score ≥ 2

Key Exclusion Criteria:

* < 18 years of age;
* pregnant or planning to become pregnant in the next 12 months;
* planned surgical or interventional procedures of the target limb (except thrombolysis and/or thrombectomy in preparation for the procedure or vena cava filter placement prior to stent implantation in patients at high risk for pulmonary embolism) within 30 days prior to or any time after the study procedure;
* planned surgical or interventional procedures for other medical conditions (i.e., not associated with the target limb) within 30 days prior to or after the study procedure;
* lesions with intended treatment lengths extending into the inferior vena cava or below the level of the lesser trochanter;
* lesion with malignant obstruction;
* previous stenting of the target vessel;
* iliofemoral venous segment unsuitable for treatment with available sizes of study devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. Comerota, MD, FACS, FACC, Principal Investigator — Inova Vascular; Lawrence "Rusty" Hofmann, MD, Principal Investigator — Stanford University
Locations (30):
- United States (29):
  - University of Alabama Birmingham Hospital, Birmingham, Alabama
  - Arrowhead Hospital, Glendale, Arizona
  - Littleton Adventist Hospital, Littleton, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Southern Connecticut Vascular Center - Norwalk Hospital, Norwalk, Connecticut
  - Christiana Care Health Systems, Newark, Delaware
  - Florida Pepin Heart Institute, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - St. Vincent Medical Group, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Louisville - Norton Hospital, Louisville, Kentucky
  - Shady Grove Adventist, Rockville, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Barnes Jewish Hospital Plaza, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - CHI Health St. Elizabeth, Lincoln, Nebraska
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York University - Langone Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - ProMedica - Jobst Vascular Institute, Toledo, Ohio
  - Oklahoma State University Medical Center, Tulsa, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Utah Valley Regional Medical Center, Provo, Utah
- Taipei Medical University Wan Fang Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hofmann LR, Gagne P, Brown JA, Saunders A, Comerota A; VIVO Study Investigators. Twelve-month end point results from the evaluation of the Zilver Vena venous stent in the treatment of symptomatic iliofemoral venous outflow obstruction (VIVO clinical study). J Vasc Surg Venous Lymphat Disord. 2023 May;11(3):532-541.e4. doi: 10.1016/j.jvsv.2022.12.066. Epub 2023 Jan 13. PMID 36646383

RESULTS

PARTICIPANT FLOW:
Groups:
- Zilver Vena Venous Self-Expanding Stent: Zilver® Vena™ Venous Stent in the treatment of symptomatic iliofemoral venous outflow obstruction.
Period: Overall Study
Arm/Group | Zilver Vena Venous Self-Expanding Stent
Started | 243
Completed | 188
Not Completed | 55
Not completed — Death | 5
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 24
Not completed — "Other" endpoint | 3

BASELINE CHARACTERISTICS:
Arm/Group | Zilver Vena Venous Self-Expanding Stent
Number analyzed (Participants) | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170
  Male | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
  Black or African American | 29
  First Nations / White | 1
  Hispanic or Latino | 7
  White | 198

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 30-day Freedom From Major Adverse Events
Description: Major adverse events were defined as procedural bleeding requiring transfusion, procedure- or device-related death, clinically driven target lesion reintervention, clinical migration, new symptomatic PE, or procedure-related perforation requiring open surgical repair or flow-limiting dissection of the target vessel.
Time Frame: 30 days
Population: The study protocol specified the analysis be based on the intent-to-treat population, which includes all 243 enrolled patients. Among the 243 enrolled patients, data for the primary safety endpoint were available for 240 patients. Therefore, because the number of analyzable patients exceeded the minimum sample size required for sufficient statistical power (n=218), the primary analysis was based on the analyzable population in accordance with the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Zilver Vena Venous Self-Expanding Stent
Number analyzed (Participants) | 240
Participants | 232
Statistical Analysis 1: Comparison: Zilver Vena Venous Self-Expanding Stent; Test type: Other; p < 0.0001, One-sided Exact binomial test; Freedom from MAE rate (%) = 96.7, 95% CI 2-sided [93.5 to 98.6] — One-sided Exact binomial test

2. Primary Outcome: The Rate of Participants With Primary Quantitative Patency at 12 Months
Description: Primary quantitative patency was defined as a treated venous segment that retained (uninterrupted; intervention-free) an MLD (Minimum Lumen Diameter ) > 50% of the immediate post-procedure stented MLD as demonstrated by venography as determined by the core laboratory.
Time Frame: 12 months
Population: The study protocol specified the primary analysis be based on intent-to-treat population (n=243). Among the 243 enrolled patients, 189 patients had venographic primary patency outcome data available (i.e., post-procedure and 12-month venogram data). Therefore, the results presented are after the outcome was imputed multiple times by random sampling from the Bernoulli distribution based on outcomes for the analyzable patients (n=189) without covariate adjustment.
Measure: Number; unit: percentage of participants
Arm/Group | Zilver Vena Venous Self-Expanding Stent
Number analyzed (Participants) | 243
percentage of participants | 89.9
Statistical Analysis 1: Comparison: Zilver Vena Venous Self-Expanding Stent; Test type: Other; p < 0.0001, Binomial test for one proportion; 12-month quantitative patency rate (%) = 89.9, 95% CI 2-sided [85.1 to 93.4] — Binomial test for one proportion

3. Secondary Outcome: Change From Baseline in the Venous Clinical Severity Score (VCSS) at 1 Month
Description: Venous Clinical Severity Score (VCSS) is a method of classifying venous disease severity based on 10 clinical descriptors (pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, number of active ulcers, duration of active ulcer, size of active ulcer, and use of compression therapy), each scored on a scale from 0 (Absent) to 3 (Severe). The VCSS score is the sum of the scores for the individual descriptors, ranging from 0 to 30.
  Mean change = (1-month score - Baseline Score)
Time Frame: Baseline and 1 month
Population: All participants with baseline and 1-month Venous Clinical Severity Score (VCSS) available. Venous Clinical Severity Score (VCSS) were available for 233 patients at 1 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zilver Vena Venous Self-Expanding Stent
Number analyzed (Participants) | 243
units on a scale
  At baseline | 8.0 (4.2)
  Change from baseline at 1 month: number analyzed (Participants) | 233
  Change from baseline at 1 month | -3.0 (0.2)
Statistical Analysis 1: Comparison: Zilver Vena Venous Self-Expanding Stent; Test type: Other; p < 0.0001, paired t-test — P-value is adjusted for multiplicity; A paired t-test with p-values adjusted for multiple comparisons using the Holm's procedure to control for a family-wise Type I error rate of 0.05; Change from Baseline Mean = -3.0, 95% CI 2-sided [-3.5 to -2.6]

4. Secondary Outcome: Change From Baseline in the Venous Clinical Severity Score (VCSS) at 12 Months
Description: Venous Clinical Severity Score (VCSS) is a method of classifying venous disease severity based on 10 clinical descriptors (pain, varicose veins, venous edema, skin pigmentation, inflammation, induration, number of active ulcers, duration of active ulcer, size of active ulcer, and use of compression therapy), each scored on a scale from 0 (Absent) to 3 (Severe). The VCSS score is the sum of the scores for the individual descriptors, ranging from 0 to 30.
  Mean change = (12-month score - Baseline Score)
Time Frame: Baseline and 12 months
Population: All participants with baseline and 12-months Venous Clinical Severity Score (VCSS) available. Venous Clinical Severity Score (VCSS) were available for 202 patients at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zilver Vena Venous Self-Expanding Stent
Number analyzed (Participants) | 243
units on a scale
  At baseline | 8.0 (4.2)
  Change from baseline at 12 months: number analyzed (Participants) | 202
  Change from baseline at 12 months | -4.2 (0.2)
Statistical Analysis 1: Comparison: Zilver Vena Venous Self-Expanding Stent; Test type: Other; p < 0.0001, pair t-test — p-value is adjusted for multiplicity; [statistical method as in outcome 3, analysis 1]; Change from Baseline Mean = -4.2, 95% CI 2-sided [-4.7 to -3.7]

ADVERSE EVENTS:
Time Frame: 3 year
Groups:
- Zilver Vena Venous Stent: Zilver Vena Venous Stent: stenting
Arm/Group | Zilver Vena Venous Stent
All-Cause Mortality (participants affected / at risk) | 5/243
Serious Adverse Events (participants affected / at risk) | 111/243
Other Adverse Events (participants affected / at risk) | 84/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilver Vena Venous Stent (N=243)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (2)
Angina pectoris (Cardiac disorders) | 2 (3)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Goiter (Endocrine disorders) | 1 (1)
Corneal degeneration (Eye disorders) | 1 (2)
Orbital haemorrhage (Eye disorders) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (8)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Rectal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 3 (3)
Hernia (General disorders) | 1 (1)
Nodule (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pelvic mass (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Surgical failure (General disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Vascular stent occlusion (General disorders) | 15 (17)
Vascular stent restenosis (General disorders) | 6 (8)
Vascular stent stenosis (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 6 (7)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Babesiosis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 5 (9)
Chronic sinusitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2)
Pelvic infection (Infections and infestations) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Post procedural infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 7 (11)
Urinary tract infection (Infections and infestations) | 2 (3)
Wound infection (Infections and infestations) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (6)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Coagulation time prolonged (Investigations) | 15 (16)
Hepatic enzyme increased (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Myastenia gravis (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 3 (3)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetic wound (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Colostomy (Surgical and medical procedures) | 1 (1)
Faecal management (Surgical and medical procedures) | 1 (1)
Metabolic surgery (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5)
Embolism (Vascular disorders) | 1 (3)
Femoral artery aneurysm (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 15 (16)
Hypertension (Vascular disorders) | 2 (2)
Iliac vein stenosis (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
May-Thurner syndrome (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (1)
Vascular wall hypertrophy (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilver Vena Venous Stent (N=243)
Peripheral swelling (General disorders) | 13 (13)
Vascular stent occlusion (General disorders) | 14 (15)
Coagulation time prolonged (Investigations) | 27 (32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (27)
Haemorrhage (Vascular disorders) | 28 (33)
Peripheral venous disease (Vascular disorders) | 19 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT01970007/Prot_SAP_000.pdf